CLINICAL TRIAL: NCT01694173
Title: Tissue Distribution of F18-FDG Labelled Autologous Bone Marrow Derived Stem Cells in Patients With Type 2 Diabetes Mellitus
Brief Title: Tissue Distribution of F18-FDG Labelled Autologous Bone Marrow Derived Stem Cells in Patients With Type 2 DM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr Vikas Sood, Ph D Student, Dept of Nuclear medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STEM CELL PGI
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus, F18-FDG labelled stem cells
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stem cell therapy - SPD artery (Experimental): Stem cells will be infused into the superior pancreaticoduodenal artery.
  Interventions: Other: Stem cell therapy- SPD artery
- Stem cell therapy - splenic artery (Active Comparator): Stem cells will be infused into the splenic artery.
  Interventions: Other: Stem cell therapy- splenic artery
- Stem cell therapy-intravenous (Active Comparator): Stem cells will be given intravenously.
  Interventions: Other: Stem cell therapy-intravenous
- Normal saline placebo -sham procedure (Placebo Comparator): Sham procedure with infusion of normal saline.
  Interventions: Other: Normal saline placebo -sham procedure

INTERVENTIONS:
Other: Stem cell therapy- SPD artery — A total of 28 patients will be enrolled and randomized to four groups of 7 patients each. 7 patients will receive stem cell infusion into the superior pancreaticoduodenal artery. Another 7 patients will be given stem cell infusion into the splenic artery. The next batch of 7 patients will receive stem cell infusion from the peripheral intravenous route and 7 patients will act as controls undergoing a sham procedure with infusion of normal saline.
  Other Names: Autologous bone marrow derived stem cells; Bone marrow mononuclear cells
  Arms: Stem cell therapy - SPD artery
Other: Stem cell therapy- splenic artery — 7 patients will receive stem cells infusion through splenic artery.
  Arms: Stem cell therapy - splenic artery
Other: Stem cell therapy-intravenous — 7 patients will receive stem cells infusion through peripheral intravenous route.
  Arms: Stem cell therapy-intravenous
Other: Normal saline placebo -sham procedure — 7 patients will receive infusion of normal saline and will act as control groups
  Arms: Normal saline placebo -sham procedure

SUMMARY:
Investigators purpose is to track stem cells in vivo in the type 2 diabetes mellitus patients after the same have been labelled with positron emission tomography tracer F18-FDG; as it is assumed that the therapeutic outcome will profoundly depend on the delivery of these cells to pancreas. Biodistribution and quantification studies will be done at 30 minutes and 90 minutes of stem cell infusion.

DETAILED DESCRIPTION:
Autologous bone marrow derived stem cells have a promising potential in regenerative medicine. In particular the past decade has garnered a great interest in cellular therapy for treating Type2 diabetes mellitus. The pertinent questions in regenerative medicine today are to know about the homing, survival, differentiation and functionality of the cells and based on these to find out the adequate administration methods and choose the optimal dose and cell types. Various modalities have been used in the preclinical and clinical trials. These include MRI,optical imaging in the form of bioluminescence and fluorescence, quantum dots, SPECT and PET/CT imaging. However the methods which are suitable for stem cell tracking in small animals are not easily translated for human trials. In humans PET/CT imaging with its reasonable resolution and unique ability to combine anatomical and functional imaging is considered to be the best bet yet. Hence we intend to label the autologous bone marrow derived stem cells with PET tracer F18-FDG and carry out biodistribution studies, our ultimate aim being to study how in vivo distribution of the cells affect therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM between 30 and 70 years of age.
* Failure to triple OHA and on stable doses of insulin for at least 3 months.
* On vildagliptin, pioglitazone and metformin for at least 3 months along with Insulin to maintain euglycemia.
* HbA1c of 6.5-7.5%
* Insulin requirement ≥0.4 IU/kg/d.
* Glutamic acid decarboxylase (GAD 65) antibody negative status.

Exclusion Criteria:

* Patients with T1DM or secondary diabetes.
* Patients with serum creatinine > 1.5 mg/dl.
* Abnormal liver function tests (defined as value of transaminases > 3 times the upper value of normal or serum bilirubin higher than normal for the reference value for the laboratory).
* History of pancreatitis
* Seropositivity for HIV, HBsAg and HCV.
* History of myocardial infarction or unstable angina in the previous 3 months.
* History of malignancy
* Patients with active infections.
* Female patients who are pregnant or lactating

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
• Increment in glucagon stimulated C - peptide levels at the end of 6 months of ABMSCT, as compared to baseline | 6 months

SECONDARY OUTCOMES:
• Any reduction in requirement of insulin dosage measured as a percentage decrease from baseline • Improvement of HbA1c levels as compared to baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bhagwant R Mittal, MBBS,DRM,MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India